CLINICAL TRIAL: NCT01464372
Title: Electrical Field Stimulation for the Treatment of Urge Urinary Incontinence and Overactive Bladder - Version: 3.0 Dated 16 APR 2012.
Brief Title: Electromagnetic Stimulation for the Treatment of Urge Urinary Incontinence and Overactive Bladder
Acronym: ELEC STIM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: EMKinetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMK0910
Record Dates: First submitted 2011-10-31; First posted 2011-11-03 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Urinary Incontinence, Urge
Keywords: Urinary Incontinence, Urge; Peripheral Nerve Stimulation
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Device (Experimental): Treatment using electrical field stimulation of peripheral nerves
  Interventions: Device: Electrical Field Stimulation Device
- Sham Device (Sham Comparator): Control group using sham device to mimic sound and sensation of investigational device
  Interventions: Device: Sham Nerve Stimulation Device

INTERVENTIONS:
Device: Electrical Field Stimulation Device — Treatment with Electrical Field Stimulation Device
  Arms: Investigational Device
Device: Sham Nerve Stimulation Device — Use of the sham device
  Arms: Sham Device

SUMMARY:
The purpose of this study is to collect data on the safety and efficacy of using an electrical field stimulation device, compared to a sham (placebo) device, to treat urinary urgency, urinary frequency and urge incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Urinary Urge Incontinence
* Urinary Frequency

Exclusion Criteria:

* Primary complaint of Stress Incontinence
* Neurogenic bladder
* Overflow Incontinence
* Functional Incontinence

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-10; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Reduction of incontinence episodes from baseline to follow-up greater for device arm than sham arm | One week after final treatment visit
  Significant increase in the percentage of patients reporting a reduction in number of incontinence episodes per day for the investigational device vs. sham
No Serious Adverse Events or Unanticipated Adverse Device Effects | First treatment through follow-up (one week after last treatment)
  Freedom from Serious Adverse Events or Unanticipated Adverse Device Effects related to procedure and/or investigational device through follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, MD, Principal Investigator — Birmingham Urologic Associates; Scott MacDiarmid, MD, Principal Investigator — Alliance Urology Specialists